CLINICAL TRIAL: NCT05417386
Title: A Phase IB Study FOLFIRINOX and NIS793 in Patients With Pancreatic Cancer
Brief Title: FOLFIRINOX + NIS793 in Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: NIS793 is no longer being developed
Sponsor: Colin D. Weekes, M.D., PhD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Colin D. Weekes, M.D., PhD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-082
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pancreas Cancer; Metastatic Pancreatic Cancer; Metastatic Pancreatic Adenocarcinoma
Keywords: Pancreas Cancer; Metastatic Pancreatic Cancer; Metastatic Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin; NIS-793; Chemoradiotherapy; Capecitabine; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-In (Experimental): Following a 3 + 3 dose escalation design 6-18 participants will receive NIS793 and FOLFIRINOX on day 1 of each 14 day cycle for 3+ cycles until recommended phase 2 dose is determined.
  Interventions: Drug: FOLFIRINOX; Drug: NIS793
- FOLFIRINOX (Experimental): Participants will be randomly assigned to receive:
  * FOLFIRINOX on day 1 of each 14 day cycle for cycles 1-8
  * Cycles 9+: Chemoradiation (CRT) and surgery
  Interventions: Drug: FOLFIRINOX; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-Fluorouracil (5-FU); Radiation: Chemoradiation; Drug: Capecitabine; Radiation: Radiation Therapy; Procedure: Surgery
- FOLFIRINOX + NIS793 (Experimental): Participants will be randomly assigned to receive:
  * FOLFIRINOX FOLFIRINOX + NIS793 on day 1 of each 14 day cycle for cycles 1-8
  * Cycles 9+: Chemoradiation (CRT) with NIS793, Surgery, NIS793
  Interventions: Drug: FOLFIRINOX; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-Fluorouracil (5-FU); Drug: NIS793; Radiation: Chemoradiation; Drug: Capecitabine; Radiation: Radiation Therapy; Procedure: Surgery

INTERVENTIONS:
Drug: FOLFIRINOX — Combination of the drugs 5-Fluorouracil (5-FU), Oxaliplatin, Irinotecan, and Leucovorin given by intravenous infusion
  Other Names: 5FU, leucovorin, irinotecan, oxaliplatin
Drug: Oxaliplatin — Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Other Names: Eloxatin
  Arms: FOLFIRINOX; FOLFIRINOX + NIS793
Drug: Leucovorin — Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Other Names: Calcium Leucovorin; Citrovorum Factor; Folinic Acid
  Arms: FOLFIRINOX; FOLFIRINOX + NIS793
Drug: Irinotecan — Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Other Names: Camptosar; Camptothecin-11; CPT-1
  Arms: FOLFIRINOX; FOLFIRINOX + NIS793
Drug: 5-Fluorouracil (5-FU) — Part of the FOLFIRINOX drug combination, given by intravenous infusion
  Other Names: Adrucil
  Arms: FOLFIRINOX; FOLFIRINOX + NIS793
Drug: NIS793 — Given by intravenous infusion
  Other Names: Nisevokitug
  Arms: FOLFIRINOX + NIS793; Safety Run-In
Radiation: Chemoradiation — Combination of Chemo (Capecitabine) and Radiation Therapy
  Arms: FOLFIRINOX; FOLFIRINOX + NIS793
Drug: Capecitabine — Taken Orally as part of Chemoradiation
  Other Names: Xeloda
  Arms: FOLFIRINOX; FOLFIRINOX + NIS793
Radiation: Radiation Therapy — Radiation Therapy as part of Chemoradiation
  Arms: FOLFIRINOX; FOLFIRINOX + NIS793
Procedure: Surgery — Surgical removal of tumor
  Arms: FOLFIRINOX; FOLFIRINOX + NIS793

SUMMARY:
This research is being done to evaluate the safety and effectiveness of the drug NIS793 in combination with the standard of care treatment FOLFIRINOX (consists of the drugs 5-Fluorouracil (5-FU), Oxaliplatin, Irinotecan, and Leucovorin), chemoradiation and surgery for people with metastatic pancreas adenocarcinoma.

The drugs involved in this study are:

* NIS793
* FOLFIRINOX (consists of the drugs 5-Fluorouracil (5-FU), Oxaliplatin, Irinotecan, and Leucovorin)

Other interventions include

* chemoradiation
* surgery.

DETAILED DESCRIPTION:
This is a two part Phase 1B study investigating whether NIS793 improves the clinical benefit of FOLFIRINOX treatment for metastatic pancreas adenocarcinoma.The first part is a safety run-in using a dose escalation strategy to determine the recommended phase 2 dose of the drug NIS793. In the second part participants will be a randomized assigned to receive either FOLFIRINOX plus NIS793 or FOLFIRINOX alone.

NIS793 binds to the protein that can be found on tumor cells, called TGFβ, thereby preventing its role in cancer metastasis (spreading). FOLFIRINOX is a combination of 4 chemotherapy drugs that may help shrink tumors.

The U.S. Food and Drug Administration (FDA) has not approved NIS793 as a treatment for any disease.

The FDA has approved FOLFIRINOX as a treatment option for metastatic pancreas adenocarcinoma The FDA has not approved the combination of NIS793 and FOLFIRINOX as a treatment for any disease.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

It is expected that about 50 people will take part in this research study.

Novartis, a pharmaceutical company, is supporting this research study by providing funding for the study, including the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Safety Run-in Cohort: Histologically confirmed metastatic pancreatic adenocarcinoma without prior therapy for pancreatic adenocarcinoma.
* Phase 1B Cohort: Histologically confirmed locally advanced disease (borderline resectable or locally advanced pancreatic adenocarcinoma) or poorly differentiated adenosquamous carcinoma includes both borderline resectable or locally advanced disease. Patients with localized pancreas adenocarcinoma cannot have received any prior therapy for borderline resectable or locally advanced pancreas adenocarcinoma
* Borderline Resectable Disease: Defined by the NCCN as tumors with venous involvement of the SMV/portal vein demonstrated tumor abutment with or without impingement and narrowing of the lumen, either tumor thrombus or encasement but with suitable vessel proximal and distal to the area of vessel involvement, allowing for safe resection or reconstruction; gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct abutment of the hepatic artery, without extension to the celiac axis; or tumor abutment of the SMA not to exceed greater than 180 degrees of the circumference of the vessel wall.Tumors involving retroperitoneal structures that can be surgically removed (i.e.kidney), will also be included.
* Locally Advanced Pancreas Adenocarcinoma: Defined by the NCCN as: Tumors of the head that have greater than 180 degrees of SMA encasement or any celiac abutment, unreconstructable SMV or portal occlusion, or aortic invasion or encasement. Tumors of the body with SMA or celiac encasement of greater than 180 degrees, unreconstructable SMV or portal occlusion, or aortic invasion. Tumors of the tail with SMA or celiac encasement of greater than 180 degrees. Irrespective of location, all tumors with evidence of nodal metastasis outside of the resection field are deemed unresectable. Participants must have measurable disease, defined as at least one lesion that measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam. See Section 12 (Measurement of Effect) for the evaluation of measurable disease.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN) if no biliary stenting has been done OR 2.0 x ULN if patient is status post biliary stenting or two downward trending values.
  * AST(SGOT)/ALT(SGPT) Safety Run-in Metastatic Disease: < 5 x institutional ULN. Locally advanced disease: ≤3 × institutional ULN
  * Creatinine ≤ institutional ULN OR
  * Glomerular filtration rate (GFR) no lower than 60 mL/min/1.73 m2

    * Creatinine clearance for males = (140 - age [yrs]) (body wt [kg]) / (72) (serum creatinine [mg/dL])
    * Creatinine clearance for females = 0.85 x male value
* Human immunodeficiency virus (HIV)-infected participants on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. Additionally, participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.

To be eligible for this trial, participants should be class. To be eligible for study participation, participants must be class 2 B or better.

* The effects of treatment on the developing human fetus are unknown. For this reason, all patients of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 9 months after completion of mFOLFIRINOX or NIS793 administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Metastatic Disease Safety Run-in: Any prior chemotherapy, radiation therapy, immunotherapy, biologic ('targeted') therapy or investigational therapy for pancreas adenocarcinoma.
* Locally Advanced Disease Cohort: Any prior chemotherapy, radiation therapy, immunotherapy, biologic ('targeted') therapy or investigational therapy for treatment of the patient's pancreatic tumor.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery
* Patients with deficient mismatch/microsatellite unstable or high tumor mutation burden cancers.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Patients requiring use of steroids to treat active uncontrolled brain metastases will be excluded from study enrollment. Patients treated with radiation > 4 weeks prior with follow up imaging showing control are eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to NIS793, 5-fluorouracil, irinotecan and oxaliplatin not amenable to institutional chemotherapy desensitization protocol.
* Known, existing uncontrolled coagulopathy. Concomitant treatment with full dose warfarin (coumadin) is NOT allowed. Patients may receive low molecular weight heparin (LMWH) (such as enoxaparin and dalteparin) and direct oral anticoagulant (DOAC) for management of deep venous thrombosis (DVT).
* History of bleeding diathesis or recent major bleeding events (i.e. Grade > 2 bleeding events in the month prior to treatment).
* Concomitant use of cimetidine, as it can decrease clearance of 5FU. Another H2- blocker or proton pump inhibitor may be substituted before study entry.
* Patient with cardiac ventricular arrhythmias requiring antiarrhythmic therapy, or atrioventricular heart block (due to 5FU administration)
* Participants with uncontrolled intercurrent illness or infection.
* Participants with uncontrolled seizures, central nervous system disorders or psychiatric illness/social situations that would limit compliance with study requirements.
* Has received a live vaccine within 30 days of planned start of study therapy. Note:

Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed. COVID non-live vaccines are allowed.

* History of severe hypersensitivity reaction to any monoclonal antibody.
* Patient with known history of UGT1A1 gene polymorphism, Patient with known history of UGT1A1 gene polymorphism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Safety Run In-Recommended Phase 2 dose (RP2D) | Up to 2 months after baseline
  Primary endpoint of safety run-in cohort is to define the recommended phase 2 dose as analyzed by 2-dimensional imaging (Computed Tomography, CT) or MRI utilizing Response Evaluation Criteria in Solid Tumors (RECIST v.1.1), obtained at 4-cycle therapy intervals.
R0 Resection Rate | Up to 8 months after baseline
  The primary endpoint of the two-arm non-comparative phase IB study (Part 2) is to estimate the R0 resection rate associated with the FOLFIRINOX/NIS793 therapy administered as neoadjuvant therapy.

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | Up to approximately 6 years after baseline
  Defined as the time from time of surgical resection of pancreas tumor to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Progression-free survival (PFS) | Up to approximately 6 years after baseline
  Defined from the date of randomization or registration to the earliest date of progressive disease or death due to any cause. Progressive disease must be documented objectively in one or more local and/or distant sites. PFS will be censored at the date of last follow-up for patients alive without documented progression.
  PFS curves will be estimated by the Kaplan-Meier method and compared using the logrank test.
Overall survival (OS) | Up to approximately 6 years after baseline
  Defined as date of randomization or registration to the date of death due to any cause and censored at the date of last follow-up for patients still alive. OS curves will be estimated by the Kaplan-Meier method and compared using the log-rank test.
Pathologic complete response (pCR) | up to 8 months after baseline
  Defined as no residual cancer in the pancreatic tissue at surgical resection. The pCR rate will be reported among all eligible patients as well as among resected patients with 95% confidence intervals based on the exact binomial distribution. Comparisons between arms may be assessed using Fisher's exact test.
Resection rate | up to 8 months after baseline
  Percentage of patient who undergo resection of their primary tumor, regardless of microscopic location of residual tumor to location of the resection margin.

CONTACTS AND LOCATIONS:
Overall Officials: Colin D Weekes, MD, PHD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation